CLINICAL TRIAL: NCT03698682
Title: Evaluation of Two Strategies of Antibiotic Treatment With Levofloxacin in Acute Exacerbation of Chronic Obstructive Pulmonary Disease: Short Treatment-versus Standard Treatment
Brief Title: Short Compared With Standard Duration of Antibiotic Treatment for AECOPD
Acronym: AECOPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AECOPD levofloxacine Study
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short treatment group (Experimental): 1 tablet Levofloxacin 500mg / day for two days completed by 1 tablet Placebo Levofloxacin 500mg / day for 5 days.
  Interventions: Drug: Levofloxacin 500mg
- Standard treatment group (Experimental): 1 tablet of Levofloxacin 500mg prescribed for 7days
  Interventions: Drug: Levofloxacin 500mg

INTERVENTIONS:
Drug: Levofloxacin 500mg — One tablet per day for 7 days.
  Other Names: Placebo Levofloxacin 500mg

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the most common diseases in the world. Acute exacerbation of COPD (AECOPD) refers to an exaggeration of the symptoms of the disease. Currently, the 3 Anthonisen criteria appear to be most satisfactory in defining the AECOPD: The increase in the volume of sputum, the alteration of its appearance which becomes purulent and The increase in dyspnea. Our recent study, showed that administration of levofloxacin is superior to placebo in the treatment of AECOPD; it is accompanied by a substantial reduction in mortality and a significant reduction in the residence time in hospital.The choice of antibiotic to be used in this situation is challenging to the clinician who must choose between traditional antibiotics (cyclins, aminopenicillins, cotrimoxazole...) and new antimicrobial agents. Antibiotic treatment duration was not based on a strong scientific rationale. Yet at the time of the dramatic emergence of bacterial resistance, reducing the selection pressure by reducing the exposure to antibiotic should be a major issue. In addition, the decrease in costs and associated side effects reinforces the interest of short treatments.

Unfortunately, few studies with a satisfactory methodology are available in the literature. In fact, we present the rational and the interest in shortening the durations of antibiotic treatment of AECOPD by levofloxacin in patients admitted to the emergency for exacerbation of COPD and to study the epidemiology of viral and bacterial AECOPD.

DETAILED DESCRIPTION:
This study is a randomized prospective double-blind, accomplished with sealed envelopes ,with two groups :

* Group A: Short treatment duration: 1 tablet Levofloxacin 500mg / day for two days completed by 1 tablet Placebo Levofloxacin 500mg / day for the remaining 5 days.
* Group B: Standard treatment duration (control group): 1 tablet Levofloxacin 500mg / day for 7 days.

The study is conducted by recruiting AECOPD patients to collect their blood samples and sputum samples. These samples will be used for the inflammatory analyses and the study of bacterial and viral serology. The results were seized by the SPSS.20.0 software.

ELIGIBILITY:
Inclusion Criteria:

45 years or older; had a smoking history of at least 10 pack-years; had a clinical diagnosis of mild-to-severe COPD, defined as a postbronchodilator forced expiratory volume in 1 s (FEV1 ) to forced vital capacity ratio of 0·7 or lower and a postbronchodilator FEV1 of at least 30%, according to Global Initiative of Chronic Obstructive Lung Disease (GOLD).

Exclusion Criteria:

Patients were excluded if they presented one of the following conditions: clinical evidence of hemodynamic compromise with need to vasoactive drugs, Glasgow coma scale <7.20, pneumonia, previous adverse reactions to study drug, antibiotic treatment in the previous days, pregnancy or lactation, severe renal (creatinineclearance 40 mL/min) or hepatic impairment, or lung disease other than COPD that couldaffect the clinical evaluation of the treatments. Patients with active alcohol or drug abuse were also excluded.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate | 30 days after inclusion
  resolution of acute signs and symptoms of the exacerbation to baseline level (non-exacerbated state), together resolution of fever if present at study entry and no recurrences nor relapse at 30 days of follow-up.

SECONDARY OUTCOMES:
Need for additional antibiotics | 30 days after inclusion
  Patient requiring additional antibiotics. The decision to initiate new antibiotics was left to the discretion of the treating physician.
ICU admission rate | 30 days after inclusion
  Patient requiring admission in an Intensive Care Unit for respiratory deterioration
Exacerbation Free Interval (EFI) | 30 days after inclusion
  The period of time duringwhich the patient is not in exacerbation. It's the period of time between two exacerbations.
Number of reexacerbation at 12 months | Up to 12 months pas inclusion
  Number of patients readmitted for exacerbation during the 12 months following inclusion
death rate at 12 months | Up to 12 months pas inclusion
  number of death at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Professor, Study Director — Research Laboratory (LR12SP18) University of Monastir 5000 Tunisia
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: officiel site — http://www.urgencemonastir.com